CLINICAL TRIAL: NCT03740451
Title: Effects of Manual Therapy on Autonomic Nervous System's Balance, Pain and Well-being in Patients With Fibromyalgia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTonANS
Record Dates: First submitted 2018-11-06; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Fibromyalgia, Manual Therapy
Keywords: Fibromyalgia, Manual Therapy, Autonomic Nervous System, Pain, Psychological well-being
MeSH Terms: conditions — Fibromyalgia; Pain; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will be conducted where patients will be divided randomly, through the website www.random.org, in three groups: 2 of them will be the experimental group and the other one will be the control group.
Who Masked: Outcomes Assessor
Masking Description: Patients will be divided randomly into 3 groups, using the website www.random.org.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): Active mobilization of soft tissues
  Interventions: Other: Active mobilization of soft tissues
- Experimental group 2 (Experimental): Passive mobilization
  Interventions: Other: Passive mobilization
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Active mobilization of soft tissues — This study will compare the effects of joint passive mobilization with the effects of soft tissue active mobilization on heart rate variability (as an indicator of autonomous regulation), psychological well-being (measured by the Ryff scale) and pain in patients with fibromyalgia.
  Arms: Experimental group 1
Other: Passive mobilization — This study will compare the effects of joint passive mobilization with the effects of soft tissue active mobilization on heart rate variability (as an indicator of autonomous regulation), psychological well-being (measured by the Ryff scale) and pain in patients with fibromyalgia.
  Arms: Experimental group 2

SUMMARY:
Scientific literature dealing with patients with fibromyalgia conveys they suffer from an abnormal response of the autonomic nervous sýstem, where a marked sympathetic hyperactivity and a decrease in heart rate variability are emphasized. It is important to know what manual therapy techniques may manage to decrease the sympathetic activity and balance the sympathetic-vagal tone, therefore improving pain and life quality.

This study will compare the effects of joint passive mobilization with the effects of soft tissue active mobilization on heart rate variability (as an indicator of autonomous regulation), psychological well-being (measured by the Ryff scale) and pain in patients with fibromyalgia.

DETAILED DESCRIPTION:
Scientific literature dealing with patients with fibromyalgia conveys they suffer from an abnormal response of the autonomic nervous sýstem, where a marked sympathetic hyperactivity and a decrease in heart rate variability are emphasized. It is important to know what manual therapy techniques may manage to decrease the sympathetic activity and balance the sympathetic-vagal tone, therefore improving pain and life quality.

This study will compare the effects of joint passive mobilization with the effects of soft tissue active mobilization on heart rate variability (as an indicator of autonomous regulation), psychological well-being (measured by the Ryff scale) and pain in patients with fibromyalgia.

The authors expect a stronger decrease in the sympathetic nervous system activation; a greater reduction in pain, and a bigger improvement in well-being and anxiety in those patients treated with active mobilization of soft tissues than passive mobilization group.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatologic diagnosis of fibromyalgia, chronic fatigue labels, sleep disorders, recurrent cervical pain associated with fibromyalgia

Exclusion Criteria:

* Smokers, blood pressure superior to 160/100 mm/Hg, coronary artery disease, peripheral vascular disease, presence of Diabetes I or II, being pregnant, psychiatric disorder established, any trauma suffered in the last 6 months, diagnosis of osteoarthritis, consumption of caffeine, alcohol or other stimulating substance at least 24 hours before the experimental intervention, performing moderate-intense physical activity 2 hours before the experimental intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-05 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Heart rate variability | 10 minutes (before, during and after intervention)
  Heart rate variability (HRV) will be assessed as an indicator of autonomic regulation. The HRV measurement will be made through the Elite HRV application, using the value of rMSSD.

SECONDARY OUTCOMES:
Pain assessed by the numerical rating scale (NRS) | 10min (before and after intervention)
  Pain will be assessed by the numerical rating scale (NRS)
Psychological well-being | 1 week (just before intervention, 1 week after intervention)
  Psychological well-being will be assessed by the Ryff scale

IPD SHARING:
Plan to Share IPD: Undecided